CLINICAL TRIAL: NCT01268800
Title: Rapid Profiling of Bone Marrow, at Presentation and After 5 Days of Induction Therapy, a Sensitive Method for Identifying Resistant AML Clones
Brief Title: Rapid Profiling of Bone Marrow, at Presentation and After 5 Days of Induction Therapy
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Rambam Health Care Campus (Other)
Responsible Party: Sponsor
Other Study IDs: 0588-10-rmb-CTIL
Record Dates: First submitted 2010-12-30; First posted 2010-12-31 (Estimated); Last update posted 2014-05-06 (Estimated); Status verified 2014-05

CONDITIONS: AML
Keywords: AML; Induction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood bone marrow and buccal smear
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- AML induction: Adults AML patients who were referred for intensive induction therapy

SUMMARY:
Personalization of AML therapy, require a reliable mechanism for accurate characterization of patient specific leukemia phenotype and genotype. Patient's specific leukemic phenotype or in practical clinical term, patient's leukemia sensitivity to induction therapy, should best investigated in-vivo during induction. Elimination of circulating leukemic blasts from peripheral blood by day 5 was shown to discriminate between good responders with superior long term survival and poor responders with poor outcome. However, many AML patients have no circulating blasts at diagnosis and even in those who have, elimination rate of it from peripheral blood was never correlated with actual response in bone marrow.

Currently, the only available source for patient's specific leukemia profile, is the bone marrow sample at diagnosis. Since leukemic blasts are heterogeneous and come from multiple different clones, "on diagnosis" marrow consist a spectrum of chemotherapy sensitive and resistance clones. Clones may vary by their molecular abnormalities and results from "on diagnosis" marrow may overlook minor resistant but existing clones. Long term prognosis is determined by those resistant clones and though our interests should be focused into the abnormalities of these clones. Residual blasts on day 5 marrow may better represent the profile of patient's leukemic resistant clones.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of acute myeloid leukemia other than APL
* Age > 18
* Patient's considered by their physician "fit" for intensive induction therapy

Exclusion Criteria:

* Withdrawal of informed consent or inability to consent
* Previous allogeneic transplantation.
* One of the following lab values persistent from presentation to day 5:

  * Serum creatinine > 2mg/dl, Direct bilirubin > 2mg/dl
  * SGOT (AST) > x4 upper limit of normal
  * Left ventricular ejection fraction < 40% as assessed 2-D echocardiogram
  * Coagulation abnormalities (INR > 1.6, PTT > x1.5 normal range)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults (>18) AML patients
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2011-02; Primary Completion 2014-08 (Estimated)

PRIMARY OUTCOMES:
complete remission | 30-54 days
  Bone marrow blasts <5% upon recovery from induction therapy

SECONDARY OUTCOMES:
Overall survival | two years
relapse rate | two years

CONTACTS AND LOCATIONS:
Overall Officials: Yishai Ofran, MD, Principal Investigator — Rambam Health Care Campus
Locations (1):
- Rambam medical center, Haifa, Israel